CLINICAL TRIAL: NCT00915161
Title: Sustained Effects of Thoracocentesis in Mechanically Ventilated Patients: an Observational Single Centre Cohort Study
Brief Title: Sustained Effects of Thoracocentesis in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Heather House, Oxford Radcliffe Research and Development
Other Study IDs: MREC-07/H0505/197
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Pleural Effusion
Keywords: ventilation; oxygenation
MeSH Terms: conditions — Pleural Effusion; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Collections of fluid around the lung (pleural effusions) are common in patients on mechanical ventilation. Long stays on mechanical ventilation can lead to serious complications such as pneumonia and are associated with significant morbidity and mortality. The drainage of pleural effusions may lead to improvements in oxygenation making it easier to discontinue mechanical ventilation.

The purpose of this study was to examine the effects of thoracocentesis (pleural fluid drainage) on blood oxygenation over a 48 hour period to see whether the effects are sustained and therefore helpful in this discontinuation.

DETAILED DESCRIPTION:
This will be a collection of data in patients in whom it has been decided by the attending clinician that pleural drainage would be beneficial. Ultrasound will be used to confirm the presence of pleural effusion and to estimate the size of the pleural effusions and to confirm the position of the pleural drain. Data will be collected before drainage, 30 minutes after drainage and then at 4,8,12 and 24 hours after the insertion of the drain (please see also attached summary of investigations). Measurements will include arterial blood gas analysis drawn from an indwelling arterial catheter, blood pressure, pulse, respiratory rate, mixed, expired CO2 and ventilator settings. The measurements will stop either at the end of the 48 hour period or when the team caring for the patient chose to remove the drain (whichever is the first).

All measurements including the arterial blood gas analysis form part of the standard care of an ICU patient. The arterial blood gas measurements are withdrawn from an indwelling arterial catheter which is routinely in place on all ICU patients. Only the use of thoracic ultrasound by a trained ultrasonographer both before and after the procedure will be additional to the standard care of the patient. The use of Chest X-rays is at the discretion of the treating clinician and does not form part of the study protocol. Standard biochemical, microbiological and cytological tests will be performed on the pleural fluid and blood in keeping with the standard practice for pleural effusions.

The primary outcome measure is the effects of drainage on the P:F ratio. measures of dead space ventilation, A-a gradiants, ventilator settings and dynamic compliance will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation with evidence of pleural effusions on plain CXR confirmed to be large on bedside ultrasound in whom the attending clinician felt drainage would be beneficial

Exclusion Criteria:

* Coagulopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on Mechanical ventilation with evidence of pleural effusion on CXR confirmed with bedside ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The ratio of Partial pressure of oxygen to inspired concentration of oxygen (P:F ratio) | pre-procedure, 30 minutes, 4,8,24 and 48 hours post procedure

SECONDARY OUTCOMES:
Effects on A-a gradients, dead space ventilation, ventilator settings and dynamic compliance | pre-procedure, 30minutes, 4,8,24 and 48 hours post procedure

CONTACTS AND LOCATIONS:
Overall Officials: andrew p walden, PhD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe hospital, Oxford, Oxon, United Kingdom

REFERENCES:
- [Derived] Walden AP, Garrard CS, Salmon J. Sustained effects of thoracocentesis on oxygenation in mechanically ventilated patients. Respirology. 2010 Aug;15(6):986-92. doi: 10.1111/j.1440-1843.2010.01810.x. Epub 2010 Jul 20. PMID 20646244